CLINICAL TRIAL: NCT00143637
Title: Dose Response Relations for Health Effects Caused by Office Dust.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Service Branchens Arbejdsgiverforening i Danmark (Unknown)
Responsible Party: Lars Mølhave Associate prof., Aarhus University
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: FORMAS 24.2/2003-0464; DORES2002
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Discomfort Symptoms; Changed Lung Function
Keywords: Office dust; Glucan; dose-response; lung function; peak expiratory flow; inflammation; perception
MeSH Terms: conditions — Inflammation | interventions — Glucans; Environment, Controlled

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Office dust with added glucan
  Interventions: Other: Office dust
- 1 (Experimental): Clean air exposures in climate chamber
  Interventions: Other: clean air

INTERVENTIONS:
Other: Office dust — airborne office dust spiked with glucan
  Other Names: Glucan
  Arms: 2
Other: clean air — Clean air
  Arms: 1

SUMMARY:
The study is focused at the dose response relation for office dust and such office dust spiked with components from fungi known from damp buildings.

The first aim of this study is to investigate if dust causes objective changes such as changes of lung function, nasal geometry, inflammatory indicators in tears and nasal lavage, tear film stability and cells at exposure levels relevant to indoor air. The controlled exposure variable is air concentration of office dust spiked with Glucan to simulate a worse case scenario.

Aim 1: Confirm or support the causality between objective effects and exposures to dust spiked with Glucan with focus on inflammatory responses. This is done by negation of the hypothesis that no significant effects are found for the variables in question.

Aim 2 is to estimate the thresholds and slopes of the DR relation for effect measures which show effects of exposures. At best the study will supply for each variable a zero response to clean air and three non-zero responses to dust. Thresholds and slopes are estimated graphically by linear regression or by an accumulated response model.

Aim 3 is a confirmation that atopic persons and histamine sensitive persons in nasal provocation tests have different responses in the effect measures showing significant effects of exposures to dust spiked with Glucan. Risk group status is therefore included in the analyses of the main variables as explaining variable.

Potential additional aim 4: Chemical and biological characterization of the office dust used in the study.

Aim 4 is an investigation of dose response relations for explorative measures, which in previous investigations have showed indications of a dose response relation. For these no a priory hypotheses exists and the analyses must be arranged ad hoc. The explaining variables are exposure and risk group status.

One challenge in investigations of unspecific effects caused by mixed exposures is that few specific objective effects measures are available and subjective measures have to be introduced. Therefore there is a need for developments of new objective measures of health effects of air pollution. Some of these are related to new biomarkers of respiratory effects in a bio-sample taken as condensed exhaled breath.

Aim 5: Developments of new objective measures of health effects of air pollution. After the experiment it will be investigated by logistic regression if a sensitivity index can be established.

DETAILED DESCRIPTION:
The basic procedure is an exposure experiment in which human subjects are exposed to controlled variations of dust spiked with Glucan. Their responses are monitored before, after minutes and hours of exposure and later the same evening.

Two groups of subjects are selected in a pre-investigation using strict selection and exclusion criteria. The two groups are atopic persons and responders to Histamine in a RSM nasal provocation test.

The groups are exposed under controlled conditions in a climate chamber at IMA to office dust spiked with Glucan (same procedure and amount as in DAMOS) at clean air level (less than 20 micro-g/m3 (TSP) and at 150, 300 and 700 micro-g/m3 (TSP). In the pre-investigation and during the exposure sessions a number of personal characteristics are measured or registered to be used in the statistical analyses as explaining variables for the responses of the subjects.

The dust exposure will be characterized both though its size distribution and gravimetrically using up-to-date analytical instruments. To optimise the exposures several pilot studies are made. Only effects measures, which previously have shown clear indications of responses to dust exposures, are included in the study.

The timetable includes pre-investigations, two repetitions of the exposure design (run 1 and 2), analyses of the bio-samples, statistical analyses, and reporting.

The study includes a main study and several additional work-packages, which will be activated when funding become available.

ELIGIBILITY:
Inclusion Criteria:

* All in local area
* Nasal histamine responsive
* Grass allergic

Exclusion Criteria:

* Pregnancy
* House dust allergy
* Hyper-responding air ways, Disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Lung Inflammation | during exposures

SECONDARY OUTCOMES:
Lung function | during exposures
FEV | during exposures
FVC | during exposures
Acoustic rhinometry | during exposures
cytokine profile | during exposures
Peak expiratory flow | during exposures
inflammation and sensory symptoms | during exposures

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mølhave, DMSc, Ph.D., Principal Investigator — The Air Pollution Unit, Department of Environmental and Occupational Medicine, Institute of Public Health, The University of Aarhus.
Locations (1):
- The Air Pollution Unit, Department of Environmental and Occupational Medicine, Institute of Public Health, The University of Aarhus., Aarhus, Denmark